CLINICAL TRIAL: NCT02311543
Title: Impact of a Surgical Sealing Patch on Lymphatic Drainage After Axillary Lymph Node Dissection for Breast Cancer. A Multicenter Randomized Phase III Trial.
Brief Title: Impact of a Surgical Sealing Patch on Lymphatic Drainage After ALND for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SAKK 23/13
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: Axillary Lymph Node Dissection (ALND); Breast Cancer; TachoSil®; Lymphatic Drainage; Surgical Sealing Patch
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: no TachoSil® (No Intervention): After axillary lymph node dissection no surgical sealing patch (TachoSil®) is applied.
- Arm B: TachoSil® (Active Comparator): After axillary lymph node dissection, 3 large TachoSil® patches in the dissected axilla are positioned to cover as much of the axillary walls as possible.
  Interventions: Drug: TachoSil® patches

INTERVENTIONS:
Drug: TachoSil® patches — TachoSil® is a sterile, ready-to-use, absorbable surgical patch and consists of an equine collagen sponge coated with human fibrinogen and human thrombin.
  Arms: Arm B: TachoSil®

SUMMARY:
Axillary lymph node dissection remains an integral part of surgical treatment of primarily node-positive invasive breast cancer. In order to reduce the incidence of clinically relevant seroma, a suction drain is routinely placed into the axillary cavity after axillary lymph node dissection (ALND) by a separate stab incision. The pathogenesis of seroma involves the collection of lymph fluid caused by dissection of lymph vessels and exudate. All coagulation and fibrinolytic factors are produced and secreted by lymphatic endothelial cells and are involved in the sealing of lymphatic capillaries. Local hemostyptic agents may therefore reduce postoperative secretion from lymphatic fistulas caused by ALND.

We propose to conduct a multicenter prospective randomized control trial in Switzerland to evaluate the impact of TachoSil®, a ready-to-use, absorbable surgical patch (consisting of an equine collagen sponge coated with human fibrinogen and human thrombin) on axillary drainage after ALND for breast cancer. We hypothesize that the use of TachoSil® significantly and relevantly reduces the volume and duration of axillary drainage after ALND. This has the potential to increase patients' quality of life, as well as to shorten the length of hospital stay and reduce hospital costs.

DETAILED DESCRIPTION:
DISEASE BACKGROUND

In Switzerland, 5'500 women and 30 to 40 men are diagnosed with breast cancer every year. It accounts for one third of all cancer diagnoses among women, and causes approximately 1'350 deaths per year. Around 1'200 patients per year need axillary lymph node dissection (ALND) as part of their surgical treatment. ALND is indicated primarily for node-positive breast cancer. Patients are identified either by pre-operative evaluation of the axilla or by intraoperative sentinel lymph node biopsy (SLNB).

THERAPY BACKGROUND

During axillary lymph node dissection for breast cancer, standard techniques for prevention of leakage of dissected lymphatic vessels include the application of suture ligaments and the use of bipolar electrocautery. Seroma prevention after ALND is achieved by placement of a closed suction drain through the skin into the axillary cavity.

Closed axillary suction drains are archaic tools to prevent seroma after ALND by simple mechanical drainage at the cost of significant patient discomfort and increased length of hospital stay. The sealing agent TachoSil® (consists of an equine collagen sponge coated with human fibrinogen and human thrombin) allows a more nuanced approach to the management of axillary seroma prevention and may support ongoing and decades-old efforts of the professional breast cancer community to decrease the duration of axillary drainage and finally, to abandon the drain from routine clinical practice.

RATIONALE FOR PERFORMING THE TRIAL

Axillary lymph node dissection remains an integral part of surgical treatment of primarily node-positive invasive breast cancer. In order to reduce the incidence of clinically relevant seroma, a suction drain is routinely placed into the axillary cavity after ALND by a separate stab incision. Indeed, a recent meta-analysis of 6 randomized controlled trials (RCT's) on axillary drainage versus no axillary drainage and a similar meta-analysis of 6 RCT's on volume-controlled versus no/short-term drainage demonstrated a significant reduction of seroma risk with the use of axillary drainage. Importantly, however, the majority of patients in these trials did not develop seroma even in the absence of axillary drainage.

The reduction of seroma risk by axillary drainage in these trials was achieved at the expense of a prolonged hospital stay and significant patient discomfort caused by the drain. During the past 4 decades at least 50 RCT's have been performed on various interventions to reduce axillary drainage with the aim of abandoning the axillary drain from clinical practice. The interventions ranged from surgical dead space reduction, use of various surgical equipment, shoulder immobilization, compression dressing, to the application of somatostatin analogons and other medication. Due to the overall limited success of these trials axillary drainage is still standard of care after ALND.

The pathogenesis of seroma involves the collection of lymph fluid caused by dissection of lymph vessels and exudate. All coagulation and fibrinolytic factors are produced and secreted by lymphatic endothelial cells and are involved in the sealing of lymphatic capillaries. Local hemostyptic agents may therefore reduce postoperative secretion from lymphatic fistulas caused by ALND. However, the results of the trials on the use of fibrin sealant in the axillary cavity after ALND were conflicting. While some showed no favorable impact of fibrin sealant, others demonstrated promising results when using fibrin glue. Consequently, a meta-analysis of 11 RCT's with 632 patients showed no impact of the use of fibrin glues after ALND on the risk of seroma or the length of hospital stay, but revealed a trend toward less drainage volume (weighted mean difference - 117.7, 95 per cent confidence interval - 259.2 to 23.8 ml). In all these studies, however, the liquid form of fibrin sealant was used.

The use of TachoSil®, which is a non-liquid surgical patch, has been shown to strongly reduce the lymphatic drainage after lymphadenectomy in gynecologic and urologic procedures and prevented the development of chylothorax in patients who underwent heart surgery with intraoperative lymphatic leakage.

We propose to conduct a multicenter prospective RCT in Switzerland to evaluate the impact of TachoSil® on axillary drainage after ALND for breast cancer. We hypothesize that the use of TachoSil® significantly and relevantly reduces the volume and duration of axillary drainage after ALND. This has the potential to increase patients' quality of life, as well as to shorten the length of hospital stay and reduce hospital costs, and provides the rationale and the clinical relevance for the proposed RCT. If the proposed RCT shows a minimum of 33% relative drainage reduction, a follow-up trial is justified. The follow-up trial will be conducted with all patients receiving TachoSil® and randomization with versus without axillary drainage. Therefore, the final goal is the omission of axillary drainage after ALND in the future.

ELIGIBILITY:
Inclusion Criteria:

at registration

* Patient has given written informed consent before registration
* Female patients; eligible for primary ALND or sentinel lymph node procedure with frozen section and either:
* newly diagnosed
* or recurrent breast cancer in the conserved breast, chest wall or axilla
* Patients with histo- or cytology proven breast cancer UICC/AJCC stage I-III
* Age ≥ 18 years
* Fluency in either German, French, Italian, Spanish, Turkish or English
* The EQ-5D questionnaire has been completed at registration
* Patient with child-bearing potential, willing to use effective contraception, not currently pregnant and agreeing not to become pregnant after trial registration and during the 24 weeks after surgery
* A negative pregnancy test within 14 days prior to inclusion is available for all women with child-bearing potential

Inclusion criteria at randomization

- ALND indicated according to clinical standards, either as single procedure or in combination with breast conserving surgery

Exclusion Criteria at registration:

* Known hypersensitivity for TachoSil® or fibrin sealant
* Patients with mastectomy (simultaneously or within 1 month before registration); patients undergoing completion mastectomy at a later day will remain eligible and are evaluable for analysis according to intention to treat. If the axillary drain is still in place at the time of completion mastectomy and a separate drain is inserted underneath the skin flaps, only the axillary drain will be considered
* Prior axillary dissection (except prior sentinel node procedure)
* Prior axillary radiotherapy
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out QoL forms
* Concurrent treatment with other experimental drugs or treatment in a clinical trial within 30 days prior to trial entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Total volume of axillary drainage | until drain removal (2 - 10 days after surgery)
  Total volume of axillary drainage in ml until drain removal.

SECONDARY OUTCOMES:
Volume of axillary drainage per 24 hours | until drain removal (2 - 10 days after surgery)
  Volume of axillary drainage per 24 hours in ml will be calculated as the total volume of axillary drainage in ml until drain removal divided by the total duration of axillary drainage in days
Total duration of axillary drainage in days | until drain removal (2 - 10 days after surgery)
  Total duration of axillary drainage in days will be calculated from the date of surgery to the date of axillary drain removal
Duration of postoperative hospital stay in days | between 3-6 days after surgery
  Duration of postoperative hospital stay in days will be calculated from the date of surgery to the date of hospital discharge.
Patients with clinically relevant seroma | until 24 weeks after surgery
  Clinically relevant seroma is defined as either causing discomfort or requiring aspiration.
Number of clinically relevant seroma aspirations | until 24 weeks after surgery
  Number of clinically relevant seroma aspirations until 24 weeks after surgery
Total volume of all clinically relevant seroma aspirations in ml | until 24 weeks after surgery
  Total volume of all clinically relevant seroma aspirations in ml until 24 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Walter Weber, MD, Study Chair — University of Basel; Christoph Tausch, MD, Study Chair — Klinik Hirslanden, Zürich
Locations (16):
- Switzerland (16):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - CSSI Bellinzona/Lugano, Ospedale San Giovanni, Bellinzona
  - Brustzentrum, Klinik Engeried, Bern
  - Kantonsspital Graubünden, Chur
  - Spital Thurgau AG, Brustzentrum, Frauenfeld
  - Hôpitaux universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Tumor- und Brustzentrum ZeTuP St. Gallen, Sankt Gallen
  - Kantonsspital St. Gallen, Sankt Gallen
  - CHVC Hôpital de Sion, Sion
  - Kantonsspital Winterthur, Brustzentrum, Winterthur
  - Brust-Zentrum Seefeld, Zurich
  - Stadtspital Triemli, Zurich
  - UniversitätsSpital Zürich, Klinik für Gynäkologie, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weber WP, Tausch C, Hayoz S, Fehr MK, Ribi K, Hawle H, Lupatsch JE, Matter-Walstra K, Chiesa F, Dedes KJ, Berclaz G, Lelievre L, Hess T, Guth U, Pioch V, Sarlos D, Leo C, Canonica C, Gabriel N, Zeindler J, Cassoly E, Andrieu C, Soysal SD, Ruhstaller T, Fehr PM, Knauer M; Swiss Group for Clinical Cancer Research (SAKK). Impact of a Surgical Sealing Patch on Lymphatic Drainage After Axillary Dissection for Breast Cancer: The SAKK 23/13 Multicenter Randomized Phase III Trial. Ann Surg Oncol. 2018 Sep;25(9):2632-2640. doi: 10.1245/s10434-018-6556-9. Epub 2018 Jun 8. PMID 29948418